CLINICAL TRIAL: NCT05673135
Title: The Differences in Adverse Maternal and Fetal Outcomes Related to Hypertension in Obese Versus Non-obese Pregnant Women
Brief Title: The Outcomes of Hypertension in Obese Versus Non-obese Pregnant Women
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammed Khairy Ali, Assistant Professor, Assiut University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HT-pre
Record Dates: First submitted 2023-01-01; First posted 2023-01-06 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Hypertension in Pregnancy
MeSH Terms: conditions — Hypertension, Pregnancy-Induced | interventions — Antihypertensive Agents; High-Energy Shock Waves; Blood Cell Count; Body Mass Index

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-obese hypertensive pregnant women (Other)
  Interventions: Drug: Anti-Hypertensive; Radiation: Ultrasound; Radiation: Doppler ultrasound; Diagnostic Test: complete blood count; Diagnostic Test: Body mass index
- Obese hypertensive pregnant women (Other)
  Interventions: Drug: Anti-Hypertensive; Radiation: Ultrasound; Radiation: Doppler ultrasound; Diagnostic Test: complete blood count; Diagnostic Test: Body mass index

INTERVENTIONS:
Drug: Anti-Hypertensive — For control of the blood pressure
Radiation: Ultrasound — For assessment of gestational age and fetal weight
Radiation: Doppler ultrasound — Umbilical artery Doppler assessment
Diagnostic Test: complete blood count — For assessment of platelet count
Diagnostic Test: Body mass index — for assessment of maternal weight during pregnancy

SUMMARY:
Hypertensive disorders of pregnancy, include pre-existing and gestational hypertension, preeclampsia, and eclampsia, it complicates up to 10% of pregnancies and represents a significant cause of maternal and perinatal morbidity and mortality. Following the "National High Blood Pressure Education Program Working Group on High Blood Pressure in Pregnancy" recommendation is currently a systolic blood pressure (SBP) ⩾ of 140 mmHg and diastolic blood pressure (DBP) ⩾ of 90 mmHg. The diagnosis generally requires two separate measurements. Accepted across international guidelines are the following four categories: Chronic/pre-existing hypertension (Hypertension discovered preconception or prior to 20 weeks gestation), Gestational hypertension (Hypertension that appears de novo after 20 weeks gestation and normalizes after pregnancy), Preeclampsia-eclampsia (De novo hypertension after 20 weeks' gestation accompanied by proteinuria, other features of maternal organ dysfunction or uteroplacental dysfunction), Chronic/pre-existing hypertension with superimposed preeclampsia-eclampsia. Over the past 2 decades, extensive epidemiologic studies have clearly established that obesity is a major risk for gestational hypertension and preeclampsia. The risk of preeclampsia typically doubles with each 5-7 kg/m2 increase in pre-pregnancy. The mechanisms have only been partially explored; increased cytokine-mediated inflammation and oxidative stress, increased shear stress, dyslipidemia, and increased sympathetic activity1 have all been proposed as possible pathways. Few studies have examined the relationship between pre-pregnancy BMI, gestational weight gain (GWG), and the risk of preeclampsia. So, our study aims to evaluate the adverse maternal and fetal outcomes related to hypertension in obese and non-obese pregnant women.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged from 20-35 years.
2. Pregnant women from 28-30 weeks.
3. Pregnant women with a singleton pregnancy.
4. Women with chronic or gestational hypertension.
5. Women with normal baseline investigations (uncomplicated hypertension).
6. Obese women and non-obese women.

Exclusion Criteria:

1. Women with preeclampsia/eclampsia.
2. Women need urgent termination of pregnancy.
3. Women with co-morbidities such as diabetes, renal diseases, cardiac ...etc.
4. Women with confirmed fetal malformation.
5. Women who will refuse to participate.

Ages: 25 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 260 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
The rate of adverse maternal outcome related to hypertension in both groups | 3 month

CONTACTS AND LOCATIONS:
Locations (1):
- Women Health Hospital - Assiut university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided